CLINICAL TRIAL: NCT03206320
Title: Topical Lidocaine 2% Gel for Analgesia and Patient Comfort During Interscalene Brachial Plexus and Axillary Blocks: A Noninferiority Randomized Trial
Brief Title: Topical Lidocaine for Needle Insertion and Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York School of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Catherine Vandepitte, M.D., Anesthesiologist, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMBe1701
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Needle Insertion and Injection Pain
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Reference (Active Comparator)
  Interventions: Drug: Lidocaine Topical
- New (Experimental)
  Interventions: Drug: Lidocaine Topical

INTERVENTIONS:
Drug: Lidocaine Topical — Comparison of lidocaine topical gel with lidocaine infiltration and with no local anesthesia in reducing needle insertion and injection pain
  Arms: New; Reference

SUMMARY:
Skin infiltration with local anesthetic is commonly used to decrease patient discomfort during peripheral nerve blocks. Topically applied local anesthetic gel might provide analgesia while eliminating the need for additional injections. The primary objective of this study was a noninferiority comparison between the analgesia achieved with topical gel with that of skin infiltration for pain upon needle insertion and injection during administration of the interscalene brachial (ISBP) and axillary (AX) plexus blocks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand Dutch, French or English language, purpose and risks of the study, provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations
* Age >18 at the time of informed consent
* ASA I-III physical class
* Scheduled for elective shoulder or upper arm surgery requiring a preoperative interscalene brachial (ISBP) or axillary (AX) plexus block

Exclusion Criteria:

* History of an allergy or contra-indication to a local anesthetic
* Baseline neurological deficit
* Medical condition that will make it difficult to assess sensory distribution or communicate with a staff member
* Presence of preexisting coagulation disorders
* Infection at injection site
* Concomitant opioid therapy
* Recent history (<3 months) of drug or alcohol abuse
* Female subjects who are pregnant or currently breastfeeding, or who have a positive pregnancy test result at first visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Needle insertion pain | Immediately at the time the needle is inserted through the skin
  Pain rating (VAS)
Injection pain | Immediately at the end of the block
  Pain rating (VAS)

SECONDARY OUTCOMES:
Fearfulness | Just before the nerve block
  Likert scale from "1" (no fear) to "5" (very fearful)
Overall discomfort | Immediately at the end of the block
  Verbal rating scale from "0" (more comfortable/less painful than expected) to "10" (less comfortable/more painful than expected)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No